CLINICAL TRIAL: NCT02700750
Title: Relation Between Macular and RNFL Thickness Measurement and Quality Grading in OCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Ori Segal, M.D, Meir Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 294-15
Record Dates: First submitted 2016-02-21; First posted 2016-03-07 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Nerve Fiber Bundle Defect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OCT exam (Other): OCT exam No Arm No Intervention
  Interventions: Device: OCT exam

INTERVENTIONS:
Device: OCT exam — OCT exam

SUMMARY:
The investigators will enroll and scan normal eyes of healthy individuals using the Spectralis OCT. Each scan is graded on a scale of 0-40, with 0 representing the lowest quality and 40 the best possible one. Each of the participants will be scanned numerous times using this noninvasive imaging tool, while trying to get as many scans as possible of different quality. The differences in the parameters between the scans will then be recoded.

Collected data will include age, sex, subjects' refractive status, visual acuity, full slit lamp exam and the participants' OCT characteristics and measurements.

DETAILED DESCRIPTION:
The investigators will enroll and scan 200 normal eyes of 100 healthy individuals using the Spectralis OCT. Each scan is graded on a scale of 0-40, with 0 representing the lowest quality and 40 the best possible one. Each of the subjects will be scanned numerous times using this noninvasive imaging tool, while trying to get as many scans as possible of different quality. The differences in the parameters between the scans will then be recoded.

Collected data will include age, sex, subjects' refractive status, visual acuity, full slit lamp exam and the participants' OCT characteristics and measurements.

ELIGIBILITY:
Inclusion Criteria: At least 20/30 visual acuity (BCVA), refractive error less than ±6 diopters (D) spherical equivalent or 3 D of astigmatism, and normal-appearing optic nerve head and retina on dilated fundus examination.

Exclusion Criteria:

* Any history or evidence of eye disease or surgery.
* Intraocular pressure (IOP) more than 22 mm Hg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
correlation between quality grading and retinal and RNFL thickness | up to 24 months

IPD SHARING:
Plan to Share IPD: Undecided